CLINICAL TRIAL: NCT04065477
Title: Improving Time-Based Prospective Memory in TBI: A Feasibility and Dosing Study
Brief Title: Improving Time-Based Prospective Memory in TBI
Acronym: TBPM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Erica Weber, Research Scientist, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-1071-19
Record Dates: First submitted 2019-07-18; First posted 2019-08-22 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; TBI; Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Injuries

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Masking Description: Study staff conducting baseline and follow-up assessments will be blind as to which group participants are placed. Study staff conducting intervention sessions will be blind to participants' baseline and follow-up assessment performance.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The experimental group will receive treatment program designed to train strategic cognitive functions. Sessions will last 50 minutes and take place twice per week for 16 weeks.
  Interventions: Behavioral: computer-based cognitive rehabilitation (CBCR)
- Control group (No Intervention): The control group will receive no active treatment and will be treated as a "no-contact control" group.

INTERVENTIONS:
Behavioral: computer-based cognitive rehabilitation (CBCR) — Program designed to improve strategic cognitive domains (e.g., complex attention, working memory)
  Arms: Experimental

SUMMARY:
This research aims to test aspects of a computer-based cognitive rehabilitation program designed to improve thinking skills in individuals with traumatic brain injury (TBI).

DETAILED DESCRIPTION:
This research aims to test aspects of a computer-based cognitive rehabilitation program designed to improve thinking skills in individuals with traumatic brain injury (TBI), particularly improving the ability to remember to do things in the future.

ELIGIBILITY:
Inclusion Criteria:

* Sustained a moderate-to-severe TBI at least one year prior to assessment
* Fluent in English
* Demonstrate impairment in strategic cognitive abilities

Exclusion Criteria:

* Significant neurological history other than TBI
* Significant psychiatric history (e.g., bipolar disorder, schizophrenia)
* Significant substance abuse history
* Steroid and/or benzodiazepine use

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Intervention Tolerability Assessment Scale | baseline through final follow-up assessment (16 weeks)
  visual analog scale to assess participants' tolerability of intervention
Recruitment rate percentage | phone screen to in-person screen (within 2 weeks)
  percentage of interested participants who met eligibility criteria via phone screen are eligible at in person screen
Retention rate percentage | baseline to mid-intervention assessment #2 (8 weeks), mid-intervention assessment #3 (12 weeks), and final follow-up (16 weeks)
  adherence rate to treatment sessions within 8 weeks (i.e., attendance at 16 sessions), 12 weeks (24 sessions), and 16 weeks (32 sessions)

SECONDARY OUTCOMES:
Changes in time monitoring & time-based prospective memory | 16 weeks
  Via a task that simultaneously assesses time monitoring frequency as it relates to time-based prospective memory performance.
Changes in strategic cognitive functions (performance on NIH EXAMINER) | 16 weeks
  Via the NIH EXAMINER, a comprehensive computerized battery of tests designed to assess strategic cognitive functioning, particularly related to executive functions and related domains.

CONTACTS AND LOCATIONS:
Overall Officials: Erica Weber, PhD, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, East Hanover, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No